CLINICAL TRIAL: NCT00355095
Title: Double Blind, Placebo-controlled Study to Determine the Safety and Efficacy of Erythropoietin as an add-on Therapy of Methylprednisolone in Subjects With Acute Optic Neuritis (VISION PROTECT)
Brief Title: Safety and Efficacy Study of Erythropoietin as add-on Therapy of Methylprednisolone to Treat Acute Optic Neuritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut fuer anwendungsorientierte Forschung und klinische Studien GmbH (Other)
Responsible Party: Dirk Simon, Institut fuer anwendungsorientierte Forschung und klinische Studien gGmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0026
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Optic Neuritis
Keywords: multiple sclerosis; add-on Therapy; erythropoietin; methylprednisolone; autoimmune optic neuritis
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): erythropoietin
  Interventions: Drug: Erythropoietin
- 2 (No Intervention): Placebo

INTERVENTIONS:
Drug: Erythropoietin — intravenous daily 3.3 *10^4 Units, duration 3 days
  Other Names: Erypo®
  Arms: 1

SUMMARY:
The purpose of this study is to determine the safety and efficacy of erythropoietin as an add-on therapy to methylprednisolone in subjects with acute autoimmune optic neuritis.

DETAILED DESCRIPTION:
SUMMARY This study is a multicenter, double-blind, placebo-controlled, parallel-group study to determine the safety and efficacy of erythropoietin (Epo) as an add-on therapy to methylprednisolone (Mpred) in subjects with acute autoimmune optic neuritis.

The primary study endpoint is nerve fiber loss in the optical nerve head determined by optical coherence tomography at weeks 4, 8, and 16 compared to baseline.

Further study objectives include visual acuity, visual field perception, optic nerve atrophy determined by magnetic resonance imaging (MRI), and recovery of visual evoked potentials (VEPs).

A number of 40 subjects will be randomized in equal numbers into one of the two treatment groups.

Treatment groups:

Epo or placebo will be administered i.v. at three consecutive days. Epo or placebo is to be given once daily following application of Mpred preferably between 8 and 10 a.m..

Subjects will be randomized to one of the following two treatment groups and dosed as follows:

* Mpred at a dose of 1000 mg per day on days 1 - 3 given as an i.v. infusion AND 3.3 x 10^4 IU recombinant human Epo per day on days 1- 3 given as an i.v. bolus injection.
* Mpred at a dose of 1000 mg per day on days 1 - 3 given as an i.v. infusion AND placebo (normal saline) on days 1 - 3 given as an i.v. bolus injection.

Men and women between the ages of 18 and 50, inclusive, diagnosed with acute unilateral optic neuritis with or without prior diagnosis of multiple sclerosis (according to McDonald criteria; Polman et al., 2005) will be considered for inclusion into the study. Those subjects must have a decreased visual acuity on the affected eye to 0.5 or less and must have signed written informed consent. While safety will be monitored during the study, an efficacy evaluation will be done after all subjects have completed week 16.

Each subject included in the study will be seen by a treating neurologist and an examining neurologist as well as by an examining ophthalmologist. The treating neurologist will function as the primary treating physician and conduct all subject safety assessments. The examining ophthalmologist and the examining neurologist will conduct all evaluations of vision/optical nerve head atrophy and neurological symptoms, respectively, but will not be involved in any other aspect of patient care. A neurophysiologist will perform measurements of VEPs. MRIs will be performed by a neuroradiologist.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, candidates must meet the following eligibility criteria at the time of randomization:

* Must give written informed consent and authorize the release and use of protected health information (PHI).
* Must be 18 to 50 years old, inclusive, at the time of informed consent.
* Must have acute unilateral optic neuritis with or without prior diagnosis of MS (according to McDonald criteria).
* Symptoms related to optic neuritis must exist for no longer than 10 days prior to inclusion.
* Must have had normal visual acuity on both eyes before and no history of optic neuritis.
* Must have a decreased visual acuity on the affected eye to 0.5 or less at screening.

Exclusion Criteria:

Candidates will be excluded from study if any of the following exclusion criteria exist at the time of randomization:

Medical history:

* Abnormal laboratory results or clinical signs indicative of any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neurological (other than MS), and/or other major disease.
* History of prior optic neuritis on the affected or non-affected eye.
* History of squint or amblyopia on either side.
* Hyperopia > 3dptr on either side.
* Myopia < -5dptr on either side.
* Astigmatism > 2dptr on either side.
* Horizontal cup disc ratio > 0.5 on either side.
* Retinal nerve fiber layer thickness outside normal values (with respect to the OCT data base).
* Ocular diseases effecting visual acuity or visual fields (cataract, glaucoma, maculadegeneration, diabetic retinopathy, retinal heredodegeneration or others).
* History of elevated blood pressure.
* Systolic blood pressure of > 159 mmHg, diastolic blood pressure > 99 mmHg at screening examination.
* History of thromboembolic events.
* Frequent thromboembolic events in 1st grade family members.
* Significant surgery within the 4 weeks prior to randomization.
* History of severe allergic or anaphylactic reactions after administration of Epo.
* History of malignancy.
* History of seizures.
* Tuberculosis with ongoing or unknown activity.
* Acute gastrointestinal ulceration within the last three months.
* Acute virus, bacterial or fungus infection.
* Infection with HIV, HBV, or HCV.
* History of colitis ulcerosa, diverticulitis, or acute enteroanastomosis.
* Severe osteoporosis.
* Active immunization within 2 weeks prior to inclusion.
* Diagnosis of phenylketonuria.
* Implanted cardiac pacemaker or other non MRI-compatible metallic body implants.
* History of drug or alcohol abuse (as defined by the investigator) within 2 years prior to randomization.
* Any of the following abnormal blood tests at screening: alanine transaminase/serum glutamate-pyruvate transaminase (AST/SGPT), or aspartate transaminase/serum glutamicoxaloacetic transaminase (AST/SGOT), gamma-glutamyl-transferase (GGT), or serum creatinine > 2 times the upper limit of normal; hematocrit > the upper limit of normal.

Treatment history

* Prior treatment with cyclosporine, mitoxantrone, methotrexate, cyclophosphamide or other immunosuppressive agents.
* Treatment with corticosteroids or Epo within 30 days prior to randomization. Miscellaneous
* Female subjects considering becoming pregnant while in the study.
* Female subjects who are currently pregnant or breast-feeding.
* Previous participation in this study or any other investigational drug study within the last four weeks.
* Current enrollment in any other investigational drug study.
* Unwillingness or inability to comply with the requirements of the protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol.
* Any other reasons that, in the opinion of the investigator, the subject is determined to be unsuitable for enrollment in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
nerve fiber loss in the optical nerve head determined by optical coherence tomography at weeks 4,8 and 16 compared to baseline. Measurements at baseline and week 16 are used to calculate estimates for changes and differences between the groups. | 4 months

SECONDARY OUTCOMES:
Visual acuity and visual field perception determined at weeks 1, 4, 8, 16 compared to baseline (week 0). MRI measurements of optic nerve atrophy performed at weeks 4, 8 and 16 compared to baseline (week 0) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricarda Diem, MD Prof., Study Director — Department of Neurology University Homborg Hospital of the Saarland, Germany
Locations (3):
- Germany (3):
  - University Hospital of Hamburg-Eppendorf (Institut of Neuroimmunology and Clinical MS Research (INIMS)), Hamburg, Hamburg
  - Department of Neurology University Hospital Goettingen, Göttingen, Lower Saxony
  - Department of Neurology University Homborg Hospital of the Saarland, Germany, Homburg, Saarland

REFERENCES:
- [Background] Maier K, Rau CR, Storch MK, Sattler MB, Demmer I, Weissert R, Taheri N, Kuhnert AV, Bahr M, Diem R. Ciliary neurotrophic factor protects retinal ganglion cells from secondary cell death during acute autoimmune optic neuritis in rats. Brain Pathol. 2004 Oct;14(4):378-87. doi: 10.1111/j.1750-3639.2004.tb00081.x. PMID 15605985
- [Derived] Suhs KW, Papanagiotou P, Hein K, Pul R, Scholz K, Heesen C, Diem R. Disease Activity and Conversion into Multiple Sclerosis after Optic Neuritis Is Treated with Erythropoietin. Int J Mol Sci. 2016 Sep 30;17(10):1666. doi: 10.3390/ijms17101666. PMID 27706045
- [Derived] Suhs KW, Hein K, Sattler MB, Gorlitz A, Ciupka C, Scholz K, Kasmann-Kellner B, Papanagiotou P, Schaffler N, Restemeyer C, Bittersohl D, Hassenstein A, Seitz B, Reith W, Fassbender K, Hilgers R, Heesen C, Bahr M, Diem R. A randomized, double-blind, phase 2 study of erythropoietin in optic neuritis. Ann Neurol. 2012 Aug;72(2):199-210. doi: 10.1002/ana.23573. PMID 22926853